CLINICAL TRIAL: NCT07057921
Title: The Learning Curve of Video Laryngeal Mask Airway (Video-LMA) Use in Airway Management by Anesthesiology Residents: A Prospective Observational Study
Brief Title: The Learning Curve of Video Laryngeal Mask Airway (Video-LMA) Use in Airway Management by Anesthesiology Residents
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: GOKAEK 2025/11/22
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Laryngeal Mask Airways; Airway Devices
Keywords: Third generation supraglottic airway devices; Cumulative Sum learning curves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group Video LMA: Anesthesiology residents in training who practice the application of video LMA.

SUMMARY:
Supraglottic airway devices hold a significant role in modern airway management, and laryngeal mask airway (LMA) devices are widely utilized in clinical anesthesia practice. Recently developed video-assisted LMA systems enable direct visual assessment of device placement and positioning. This technology not only has the potential to enhance patient safety but also offers an opportunity to optimize the learning process by providing visual feedback during training.

Enhancing the technical proficiency of anesthesia residents in airway management is a fundamental component of their education. However, the contribution of next-generation devices such as video LMAs to the learning process and the characterization of their learning curve have been scarcely addressed in the literature. In this context, a quantitative evaluation of the acquisition process of video-assisted LMA insertion skills may provide valuable insights for both educational strategies and patient safety.

DETAILED DESCRIPTION:
Supraglottic airway devices constitute a fundamental component of modern airway management, with laryngeal mask airway (LMA) devices being widely implemented across various clinical anesthesia settings. The advent of video-assisted LMA systems has enabled real-time visual confirmation of device insertion and positioning, thereby enhancing procedural accuracy. Beyond their potential to improve patient safety outcomes, these advanced systems provide a pedagogical advantage by facilitating visual feedback during training, thus supporting the optimization of skill acquisition and educational effectiveness in airway management.

The primary aim of this study is to evaluate the learning curve of anesthesia residents during the placement of video-assisted laryngeal mask airway (video LMA) devices and to objectively assess our routinely implemented training protocol by systematically recording the process. Video-assisted airway devices, particularly video LMA systems, offer several advantages over conventional blind techniques. These advantages include higher success rates of insertion, shorter placement times, direct visual confirmation of proper positioning, and a reduction in airway-related complications. Today, many experts acknowledge that video-assisted techniques represent a new standard in supraglottic airway management with respect to both patient safety and educational utility.

Successful execution of video LMA placement requires the acquisition of three core and interrelated technical skills: obtaining an adequate view during insertion, correctly interpreting the visual information to assess device position, and performing precise manipulation through hand-eye coordination. These competencies are especially crucial for anesthesia residents undergoing training and must be effectively acquired during their educational development.

The use of LMA is common in routine elective surgeries. Video-assisted LMA systems are particularly beneficial in educational settings, as they provide real-time visual feedback for the operator and facilitate instructor-led guidance. Before initiating video LMA applications, residents in our institution undergo structured theoretical and practical training, followed by supervised clinical practice under the guidance of experienced anesthesiologists and academic staff. Through this study, we aim to analyze the learning curves of residents and objectively evaluate the effectiveness of the educational approach.

This study aims to evaluate the learning curves of residents in video laryngeal mask airway (LMA) placement and to objectively assess the effectiveness of the training program. This prospective observational study will be conducted with the participation of anesthesiology and reanimation residents at a university hospital. First- and second-year anesthesia residents with no prior experience in video LMA insertion will be included in the study.

Each participant will perform a predetermined number of video LMA insertions (≥10 cases) in adult patients undergoing elective surgery. For each attempt, success or failure, insertion time, quality of ventilation, and the occurrence of complications such as bleeding or gag reflex will be recorded. Success criteria will be based on standards defined in the literature, and all procedures will be carried out under the supervision of an experienced instructor.

Using the collected data, each participant's learning curve will be analyzed using the Cumulative Sum (CUSUM) method. This will allow for statistical assessment of the number of cases required for the learning process to reach a stable plateau.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiology residents with less than two years of experience and no prior exposure to video laryngeal mask airway (LMA) placement.

Exclusion Criteria:

* Having prior hands-on experience with video laryngeal mask airway (LMA) placement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Anesthesiology residents in training who practice the application of video laryngeal mask airway (video LMA).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Success rate and learning curve in the acquisition of video LMA insertion skills | From the first video LMA application attempt to the completion of the 10th attempt for each participant, within the data collection period of May 20, 2025, to August 20, 2025.
  Based on the collected data, the learning curve of each participant will be calculated using the CUSUM analysis method. This will allow a statistical evaluation of the number of cases after which the learning process stabilizes and reaches a plateau.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Selcuk Kusderci, Study Director — Samsun University
Locations (1):
- Samsun University, Samsun Training and Research Hospital, Samsun, Ilkadım, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ragazzi R, Finessi L, Farinelli I, Alvisi R, Volta CA. LMA Supreme vs i-gel--a comparison of insertion success in novices. Anaesthesia. 2012 Apr;67(4):384-8. doi: 10.1111/j.1365-2044.2011.07002.x. Epub 2012 Feb 13. PMID 22329593
- [Result] Nakanishi T, Sakamoto S, Yoshimura M, Toriumi T. A learning curve of LMA(R) ProSeal insertion: a prospective analysis of cumulative sum method. J Anesth. 2020 Aug;34(4):554-560. doi: 10.1007/s00540-020-02790-y. Epub 2020 May 23. PMID 32447454
- [Result] Nakanishi T, Sakamoto S, Yoshimura M, Fujiwara K, Toriumi T. Learning curve of i-gel insertion in novices using a cumulative sum analysis. Sci Rep. 2023 May 2;13(1):7121. doi: 10.1038/s41598-023-34152-5. PMID 37130901